CLINICAL TRIAL: NCT04123158
Title: MYometrial Lesion UltrasouNd And mRi
Acronym: MYLUNAR
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, CICCARONE FRANCESCA, Medical doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2370
Record Dates: First submitted 2019-10-09; First posted 2019-10-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Sarcoma Uterus
Keywords: Ultrasound; Myoma; MRI
MeSH Terms: conditions — Myoma | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- WHITE: If no Green Card criteria is fulfilled (Negative Green Criteria), the patient will receive an annual telephone follow up for 2 years.
  Interventions: Diagnostic Test: Ultrasound
- GREEN: Patients will be assessed by a Green Card to check the eventual presence of at least one of the following clinical and/or ultrasound characteristics.
  * If one or more Green Card criteria is present (Positive Green Criteria), a dedicated clinical and ultrasound paper form will be fulfilled in order to check the presence of the criteria described in the Orange Card
  * In case of "negative Orange Criteria" (no Orange Card criteria, or only one Orange Card criteria, or only Orange clinical criteria) the patient will be scheduled for longitudinal follow up at 6, 12 and 24 months. At each follow-up visit, a transvaginal ultrasound examination will be performed (using the MYLUNAR Paper Form) and the patient will be re-evaluated according to the Orange Card. In case of "positive Orange Criteria" the patient will be triaged to MRI and surgery. Eventual treatment for the myometrial lesion during the study period will be recorded and the outcome of these patients will be described separately.
  Interventions: Diagnostic Test: Ultrasound
- ORANGE: - If at least two Orange Card criteria (including at least one ultrasound parameter) are present (Positive Orange Criteria), the patient will be examined by means of Magnetic Resonance (MRI) within 30 days and triaged to surgery (to be performed within 60 days since the enrollment in the study). A dedicated MRI paper form will be fulfilled Histology of the target myometrial lesion will be considered as the gold standard parameter.
  Interventions: Diagnostic Test: Ultrasound; Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: Ultrasound — Intervention: Diagnostic Test Ultrasound Ultrasound investigating the following characteristics: Maximum size of the lesion ≥ 8cm; Largest diameter rapid growth (Growth >30% per year); Irregular margins of the lesion; Presence of irregular cystic areas; Absence of acoustic shadow; Color Score 4; "Cooked" aspect; ]
Diagnostic Test: MRI — Diagnostic Test: MRI; MRI investigating the following carachteristics:
  TARGET LESION Maximum diameter; Borders; Signal intensity on T2WI; Heterogeneity on T2WI; Cystic alteration(s); Cystic alteration(s) borders; Hemorrhage; T2 dark" area(s); Flow voids; Signal intensity on DWI(b-1000); ADC value; ≥ 1,23 Signal intensity on contrasted images Intensity [relative to myometrium] (Hyper- / Hypo- / Iso- intense) Heterogeneity (Homogeneous / Heterogeneous) Unenhanced area(s) Presence (Present / Absent) Location (Central / None or non-central) 1 Tumour - myometrium contrast ratio on T2WI [SItumour - SImyometrium / SImyometrium]
  Groups: ORANGE

SUMMARY:
A monocentric prospective observational study aimed at assessing the accuracy of a diagnostic algorithm to pre-operatively identify uterine sarcomas..

Primary Aim:The primary outcome is to evaluate the accuracy (sensitivity/specificity) of "Positive Orange Criteria" category in predicting uterine sarcoma and STUMP in the population of patients with > 3 cm myometrial lesions.

DETAILED DESCRIPTION:
INTRODUCTION

Uterine sarcomas are rare malignant tumors arising from the mesenchymal tissues of the uterus including the endometrial stroma, uterine muscle and connective tissue. They represent 1% of female genital tract malignancies and 3-7% of all uterine malignances with a worldwide annual incidence of 1.55-1.95 per 100.000 women. Malignant mesenchimal tumors include: uterine leiomyosarcoma (LMS), endometrial stromal sarcoma (ESS), and undifferentiated uterine sarcoma (UUS), and other (eg adenosarcoma, epithelioid sarcoma, STUMP). The current WHO classification also includes a smooth muscle tumor with features that preclude an unequivocal diagnosis of leiomyosarcoma, but do not fulfill the criteria for leiomyoma, or its variants, therefore is defined as smooth uterine muscle of uncertain malignant potential (STUMP). While most STUMP patients have good outcomes, unexpected aggressive behavior can be seen in some of the tumors.

The mean age at diagnosis is approximately 60 years old. However, uterine sarcomas have been diagnosed in women as young as 20 years old . The prevalence of sarcoma in women undergoing hysterectomy or myomectomy for a myometrial mass, is approximately 0.001 percent (1 in 1000) (Parker 94), with a range from 0.005 (1 in 2000) to 0.28 percent (1 in 352). , The discrimination between benign and malignant myometrial lesions is clinically relevant to plan the optimal management (surgery versus medical treatment) and to define the most appropriate surgical approach.

However, the diagnosis of uterine sarcomas or STUMP is a challenge and no validated clinical or radiological criteria can accurately distinguish benign from malignant myometrial tumors.

In particular, data on the ultrasound features of uterine sarcomas are scarce and they are mainly based on retrospective case series. The role of CT(Computed Tomography) has generally been limited to identify extrauterine disease, including local spread within the pelvis and metastatic disease. MRI (Magnetic Resonance Imaging) )represents an accurate diagnostic imaging modality in the assessment of gynecological pathologies with high soft tissue contrast, large field-of-view and multiplanar imaging capabilities; however, no accurate diagnostic criteria have been validated to discriminate between benign and malignant myometrial lesions.

To the best of our knowledge, no large prospective studies have been carried on to assess a diagnostic algorithm to predict the malignant histology of myometrial lesions.

PURPOSES AND OBJECTIVES OF THE CLINICAL TRIAL

Primary aim:

The primary outcome is to evaluate the accuracy (sensitivity/specificity) of "Positive Orange Criteria" category in predicting uterine sarcoma and STUMP in the population of patients with > 3 cm myometrial lesions.

Secondary aims:

1. To describe the clinical history of patients with myometrial lesions, assessed on ultrasound, and conservatively managed.
2. To assess the accuracy of subjective assessment of an experienced ultrasound examiner in detecting uterine sarcomas and STUMP in women with at least one >3 cm myometrial lesion.
3. To compare clinical and ultrasound characteristics of patients with benign myometrial lesion versus those with uterine sarcomas and STUMP, histologically confirmed.
4. To compare clinical and Magnetic Resonance (MR) characteristics of patients with benign myometrial lesions versus those with uterine sarcomas and STUMP, histologically confirmed.
5. To compare the accuracy of the subjective assessment of an ultrasound examiner versus that of a MR reader in detecting uterine sarcomas and STUMP in women triaged for surgery ("Orange group").

EXPERIMENTAL DESIGN

* Type of study: Monocentric, prospective, observational study
* Setting: Department of Woman and Child Health, Fondazione Policlinico Universitario A. Gemelli, IRCSS, Roma.
* Estimated study period: Three years for the enrollment and additional two years for the completion of follow-up.

STUDY POPULATION SAMPLE SIZE

This study is dimensioned on the hypothesis that "Positive Orange criteria" category has a sensitivity of at least 90% in identify patients with uterine sarcoma and STUMP among patients with at least one >3 cm myometrial lesion, against a null hypothesis of 65% [143]. Considering the prevalence of uterine sarcoma in this population 1.55%, as per our previous experience, to demonstrate an increase in sensitivity of 25% with a 90% power and bilateral alpha error=5%, 2000 patients (with at least one ≥ 3 cm myometrial lesion) with 30 sarcomas are needed. Considering a 15% of drop-out (patients evaluated but not completing the observation), 2353 patients will be enrolled. With this number of patients, the study will have 100% power in demonstrating a similar increase in the specificity of the "Positive Orange criteria" category with an alpha error=0.05. (PASS v11)

IDENTIFICATION PARAMETERS

A myometrial lesion with the largest diameter >3 cm represents the target lesion. In case of multiple myometrial lesions with similar ultrasound morphology, the largest tumor will be selected as target lesion. In case of multiple myometrial lesions with different ultrasound morphology, the "target lesion" will be identified by the ultrasound examiner on the basis of the parameters subjectively considered suspicious for malignancy.

WITHDRAWAL PROCEDURES

The patient may choose not to take part in this study. The patient may choose to have US revaluation or surgery without enrolling in this study. The patient may choose to receive other therapy, if available. In all cases, the woman receive appropriate medical care, including treatment for bleeding, pain or other symptoms.

SUBJECT TREATMENT

All women enrolled in the study will be managed according to the following algorithm (Figure 1. Clinical and Diagnostic Algorithm).

Patients will be assessed by a Green Card (Figure 2. Green Card) to check the eventual presence of at least one of the following clinical and/or ultrasound characteristics:

* Maximum size of the lesion ≥ 5cm;
* Symptoms (abdominal and/or pelvic pain, sensation of pressure, abdominal distension, infertility (>12 months), two or more abortions;
* Largest diameter rapid growth (Growth >30% per year);
* Irregular cystic areas;
* Color Score 4.

  * If no Green Card criteria is fulfilled (Negative Green Criteria), the patient will receive an annual telephone follow up for 2 years.
  * If one or more Green Card criteria is present (Positive Green Criteria), a dedicated clinical and ultrasound paper form (Appendix 1. MYLUNAR Paper Form) will be fulfilled in order to check the presence of the criteria described in the Orange Card (Figure 3. Orange Card):
* Anamnestic and clinical characteristics:

  * Age ≥ 45 years old
  * Symptoms (abnormal uterine bleeding; abdominal and/or pelvic pain; sensation of pressure; Abdominal distension)
  * LDH (Lactate dehydrogenase) > 250 UI/L (if known)
* Ultrasound characteristics:

  * Maximum size of the lesion ≥ 8cm
  * Largest diameter rapid growth (Growth >30% per year)
  * Irregular margins of the lesion
  * Presence of irregular cystic areas
  * Absence of acoustic shadow
  * Color Score 4
  * "Cooked" aspect

    * If at least two Orange Card criteria (including at least one ultrasound parameter) are present (Positive Orange Criteria), the patient will be examined by means of Magnetic Resonance (MRI) within 30 days and triaged to surgery (to be performed within 60 days since the enrollment in the study). A dedicated MRI paper form will be fulfilled (Appendix 2. MRI Paper Form) Histology of the target myometrial lesion will be considered as the gold standard parameter.
    * In case of "negative Orange Criteria" (i.e. no Orange Card criteria, or only one Orange Card criteria, or only Orange clinical criteria) the patient will be scheduled for longitudinal follow up at 6, 12 and 24 months. At each follow-up visit, a transvaginal ultrasound examination will be performed (using the MYLUNAR Paper Form) and the patient will be re-evaluated according to the Orange Card. In case of "positive Orange Criteria" the patient will be triaged to MRI and surgery. Eventual treatment for the myometrial lesion during the study period will be recorded and the outcome of these patients will be described separately.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to our Department for transvaginal ultrasound examination, in whom a myometrial lesion > 3cm in size is detected.
* Informed consent form signed by the patient.

Exclusion Criteria:

* Patients undergoing medical treatment for myometrial lesion;
* Patients previously treated with hormonal therapy including estroprogestin in the last six months;
* Patients previously treated by embolization

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a myometrial lesion with the largest diameter >3 cm that represents the target lesion
Sampling Method: Probability Sample
Enrollment: 2353 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic algorithm in predicting uterine sarcoma and STUMP | January 2019- January 2024
  the accuracy (sensitivity/specificity) of "Positive Orange Criteria" category in predicting uterine sarcoma and STUMP in the population of patients with > 3 cm myometrial lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Ciccarone, M.D., Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Denschlag D, Thiel FC, Ackermann S, Harter P, Juhasz-Boess I, Mallmann P, Strauss HG, Ulrich U, Horn LC, Schmidt D, Vordermark D, Vogl T, Reichardt P, Gass P, Gebhardt M, Beckmann MW. Sarcoma of the Uterus. Guideline of the DGGG (S2k-Level, AWMF Registry No. 015/074, August 2015). Geburtshilfe Frauenheilkd. 2015 Oct;75(10):1028-1042. doi: 10.1055/s-0035-1558120. Erratum In: Geburtshilfe Frauenheilkd. 2015 Oct;75(10):e3. doi: 10.1055/s-0035-1558288. PMID 26640293
- [Background] Pritts EA, Vanness DJ, Berek JS, Parker W, Feinberg R, Feinberg J, Olive DL. The prevalence of occult leiomyosarcoma at surgery for presumed uterine fibroids: a meta-analysis. Gynecol Surg. 2015;12(3):165-177. doi: 10.1007/s10397-015-0894-4. Epub 2015 May 19. PMID 26283890
- [Background] Mahnert N, Morgan D, Campbell D, Johnston C, As-Sanie S. Unexpected gynecologic malignancy diagnosed after hysterectomy performed for benign indications. Obstet Gynecol. 2015 Feb;125(2):397-405. doi: 10.1097/AOG.0000000000000642. PMID 25569001
- [Background] Norris HJ, Taylor HB. Mesenchymal tumors of the uterus. I. A clinical and pathological study of 53 endometrial stromal tumors. Cancer. 1966 Jun;19(6):755-66. doi: 10.1002/1097-0142(196606)19:63.0.co;2-u. No abstract available. PMID 5939046
- [Result] Koh WJ, Greer BE, Abu-Rustum NR, Apte SM, Campos SM, Cho KR, Chu C, Cohn D, Crispens MA, Dizon DS, Dorigo O, Eifel PJ, Fisher CM, Frederick P, Gaffney DK, George S, Han E, Higgins S, Huh WK, Lurain JR 3rd, Mariani A, Mutch D, Fader AN, Remmenga SW, Reynolds RK, Tillmanns T, Valea FA, Yashar CM, McMillian NR, Scavone JL; National Comprehensive Cancer Network. Uterine Sarcoma, Version 1.2016: Featured Updates to the NCCN Guidelines. J Natl Compr Canc Netw. 2015 Nov;13(11):1321-31. doi: 10.6004/jnccn.2015.0162. PMID 26553763